CLINICAL TRIAL: NCT06968065
Title: Comparison of Ultrasound-Guided Serratus Combination Plane Blocks and Local Wound Infiltration for Postoperative Analgesia Management in Minimally Invasive Cardiac Surgery (MICS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: İstanbul Yeni Yüzyıl Üniversitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024101338
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Pain, Postoperative; Heart Surgery; Analgesia
Keywords: Pain, Postoperative; Heart Surgery, Minimally Invasive; Analgesia; Bupivacaine; Opioid-Related Disorders
MeSH Terms: conditions — Pain, Postoperative; Agnosia; Opioid-Related Disorders | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAP + SIP Block Group (Experimental): Participants in this arm will receive a combination of ultrasound-guided serratus anterior plane (SAP) block and serratus-intercostal interfascial plane (SIP) block. The SAP block will be performed using 30 mL of 0.25% bupivacaine, and the SIP block will use 10 mL of 0.25% bupivacaine. Both blocks will be administered after surgery but before emergence from anesthesia.
  Interventions: Procedure: Ultrasound-guided serratus anterior plane block and serratus-intercostal interfascial plane block with bupivacaine
- Local Wound Infiltration Group (Active Comparator): Participants in this arm will receive local wound infiltration (LWI) consisting of 40 mL of 0.25% bupivacaine. The infiltration will be applied to the surgical and drain sites after surgery.
  Interventions: Procedure: Local wound infiltration with bupivacaine

INTERVENTIONS:
Procedure: Ultrasound-guided serratus anterior plane block and serratus-intercostal interfascial plane block with bupivacaine — Participants will receive an ultrasound-guided serratus anterior plane (SAP) block using 30 mL of 0.25% bupivacaine combined with a serratus-intercostal interfascial plane (SIP) block using 10 mL of 0.25% bupivacaine. Both blocks will be administered after surgery but before emergence from anesthesia. This combination targets multiple interfascial planes to enhance postoperative analgesia in patients undergoing minimally invasive cardiac surgery (MICS).
  Arms: SAP + SIP Block Group
Procedure: Local wound infiltration with bupivacaine — Participants will receive local wound infiltration with 40 mL of 0.25% bupivacaine applied to the surgical and drain sites following surgery. This approach represents a standard method for managing postoperative pain in MICS patients and serves as the active comparator.
  Arms: Local Wound Infiltration Group

SUMMARY:
This randomized, prospective, single-blinded study aims to compare the efficacy of ultrasound-guided serratus anterior plane (SAP) block combined with serratus-intercostal interfascial plane (SIP) block versus local wound infiltration (LWI) for postoperative analgesia in patients undergoing minimally invasive cardiac surgery (MICS). The primary outcome is total perioperative and postoperative opioid consumption. Secondary outcomes include postoperative pain scores (NRS), opioid-related side effects, block-related complications, and ICU stay duration.

DETAILED DESCRIPTION:
Minimally invasive cardiac surgery (MICS) has gained popularity due to reduced surgical trauma and faster recovery. However, postoperative pain management remains a challenge. This study evaluates the analgesic effectiveness of combining two interfascial plane blocks-SAP and SIP-under ultrasound guidance, compared to traditional local wound infiltration. A total of 60 patients scheduled for MICS with cardiopulmonary bypass will be randomized into two groups (SAP+SIP vs LWI). Pain scores, opioid usage, and complications will be recorded at predetermined intervals up to 72 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Undergoing MICS with left-sided 4th-5th intercostal incision
* ASA I-III
* Informed consent provided

Exclusion Criteria:

* Coagulopathy or on anticoagulants

  * Allergy to local anesthetics or opioids
  * Local infection at block site
  * Pregnancy or lactation
  * Bilateral thoracic incisions
  * Refusal to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
o Total opioid consumption (mcg of fentanyl and mg of tramadol) in the first 48 hours postoperatively. | 48 hours
  The cumulative perioperative and postoperative opioid consumption measured in micrograms of fentanyl and milligrams of tramadol administered during the first 48 hours after surgery.

SECONDARY OUTCOMES:
NRS pain scores (static and dynamic) at 0, 2, 4, 8, 16, 24, 48, and 72 hours postoperatively. | 0 to 72 hours postoperatively.
  Pain intensity will be assessed using the Numeric Rating Scale (NRS) at rest and during movement at predefined postoperative time points (0, 2, 4, 8, 16, 24, 48, and 72 hours).

CONTACTS AND LOCATIONS:
Locations (1):
- Kolan International Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No